CLINICAL TRIAL: NCT05753319
Title: Physiotherapist in the Emergency Department : What Impact Does the Intervention of the Physiotherapist Have on the Care Pathway of the Elderly Person Who Falls?
Brief Title: Physiotherapist in the Emergency Department
Acronym: KiUrge
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Laboratoire Motricité, Interactions, Performance (UR 4334) of Nantes University (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC23_0068
Record Dates: First submitted 2023-02-10; First posted 2023-03-03 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Emergencies; Fall
Keywords: Emergency department; Elderly person; Physiotherapist; Fall
MeSH Terms: conditions — Emergencies | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physiotherapy group: Intervention group with assessment and early physiotherapy
  Interventions: Other: Physiotherapy in the emergency department after a fall
- Control group: control group without assessment and physiotherapy in the emergency department

INTERVENTIONS:
Other: Physiotherapy in the emergency department after a fall — Realization of a physiotherapy assessment.
  Groups: Physiotherapy group

SUMMARY:
This study aims to evaluate the impact of assessment and early physiotherapy management on the care pathway of the elderly person who falls, their length of stay in hospital and their fall recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 75 and over
2. Patients admitted to emergency for falls.
3. Clinically stable patient who may benefit from a gait assessment or fall risk assessment
4. Patients able to understand the protocol and not verbally object to participation.

Exclusion Criteria:

1. Patients with limb fractures requiring surgical treatment
2. Patients under guardianship or curatorship.
3. Patients already included in an interventional research protocol.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: People aged 75 and over admitted to emergency for falls
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Patient orientation (return home, short-term hospitalization unit, hospitalization) at discharge from the emergency department | up to 48 hours
  The orientation of the patient on discharge from the emergency services, according to the three defined pathways (return home, short-term hospitalization unit, hospitalization).

SECONDARY OUTCOMES:
Length of stay in emergency departments and in the short stay hospital unit | up to 48 hours
  Calculation of the duration in hours by recording the dates and times of admission and discharge from the service.
Total duration of hospitalization for each stay, all services combined | 1 week
  Calculation of the duration in hours by recording the dates and times of admission to the emergency services and final discharge from the hospital.
Number of recurrence of emergency admission for the same reason (fall) | up to 9 days
  Recurrence of a fall within seven days of returning home
Satisfaction of doctors in emergency services | 0 day
  A satisfaction questionnaire will be sent to all doctors who participated in the study
Emergency discharge referral before and after assessment by the physical therapist. | up to 48 hours
  For the "Physiotherapy group" : Description of changes in physician orientation decision (return home, acute care unit, hospitalization) of patients, before/after the physical therapist assessment

CONTACTS AND LOCATIONS:
Overall Officials: Marie Blandin, Principal Investigator — Nantes University Hospital; Marie Gallet, Principal Investigator — marie.gallet@chu-nantes.fr; Guillaume LE SANT, PhD, Principal Investigator — Laboratoire Motricité, Interactions, Performance (UR 4334)
Locations (1):
- University Hospital of Nantes, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blandin M, Gallet M, Volteau C, Le Conte P, Rulleau T, Le Sant G. Effects of the delivery of physiotherapy on the treatment course of elderly fallers presenting to the emergency department: Protocol for a randomized clinical trial. PLoS One. 2024 May 8;19(5):e0303362. doi: 10.1371/journal.pone.0303362. eCollection 2024. PMID 38718002